CLINICAL TRIAL: NCT06587581
Title: Effectiveness of Text Messaging Intervention to Improve Dietary Behaviors Among Patients with Type 2 Diabetes Mellitus in Low Resource Area of Sabah: a Randomized, Open-Label, Controlled Trial
Brief Title: Effectiveness of Text Messaging Intervention to Improve Dietary Behaviors Among Patients with Type 2 Diabetes Mellitus in Low Resource Area of Sabah (DTEXT-SBH)
Acronym: DTEXT-SBH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Malaysia Sabah (Other)
Responsible Party: Principal Investigator, ESTHER ALIM ALBERT, REGISTERED DIETITIAN, Universiti Malaysia Sabah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RSCH ID-24-01119-NHX
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Type 2 Diabetes Mellitus(T2DM)
Keywords: type 2 diabetes mellitus; lack access to dietitian; eHealth; Dietary adherence; low resource area
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- T2DM Medical Nutrition Therapy (Active Comparator): Participants from control groups will receive the usual care, which will be a three-monthly nutrition consultation by a visiting dietitian
  Interventions: Other: Control Group
- T2DM Medical Nutrition Therapy and Text Messages (Experimental): Participants from the intervention group will receive the usual care and an additional three text messages per week via WhatsApp over the 6-month intervention period
  Interventions: Other: Intervention Group

INTERVENTIONS:
Other: Control Group — Participants from the intervention group will receive the usual care over the 6-month intervention period
  Arms: T2DM Medical Nutrition Therapy
Other: Intervention Group — Participants from the intervention group will receive the usual care and an additional three text messages per week via WhatsApp over the 6-month intervention period
  Arms: T2DM Medical Nutrition Therapy and Text Messages

SUMMARY:
The goal of this clinical trial is to learn if sending three (3) text messages per week over a six (6) months period to people with Type 2 Diabetes in areas with lack access to dietitian could help them stick to a healthier diet. The main questions it aims to answer are:

* Does a mobile phone text-message intervention improve dietary adherence among T2DM patients?
* Does a mobile phone text-message intervention improve HbA1c and self-management among T2DM patients? Researchers will compare dietary adherence, HbA1c changes and self-management behaviors between the usual care group and intervention group.

Participants will:

* Be given three (3) text messages per week over a six (6) months period for the intervention group
* Both usual care and intervention group will be given standard medical nutrition therapy at baseline, 3rd and 6th months visits to the clinic

ELIGIBILITY:
Inclusion Criteria:

* have type 2 diabetes.
* own a mobile phone.
* able to use WhatsApp.
* able to read and speak Bahasa Malaysia.
* have an HbA1c level above 7.0%.
* have not seen a dietitian in the previous 6 months.

Exclusion Criteria:

* individuals with type 1 diabetes mellitus and gestational diabetes mellitus.
* patients with cognitive impairment affecting memory, attention, language, and problem-solving skills.
* those with advanced diabetic complications, such as kidney failure and neuropathy.
* individuals lacking regular access to a mobile phone or with poor network connectivity.
* pregnant individuals or those planning to get pregnant in the next 6 months, as well as those currently nursing.
* individuals with major illnesses like cancer or advanced heart disease.
* those planning major surgery or gastric bypass in the next 6 months.
* institutionalized individuals, such as those in nursing homes, old folks' homes, or imprisoned.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Comparison of dietary adherence at 3-month and 6-month between the usual care group and intervention group | Baseline, 3-month, and 6-month
  Dietary adherence to diabetic diet will be evaluated against a modified healthy eating index (HEI). A 3-day dietary record methodology (2 weekdays and 1 weekend) will be used and analyzed based on Malaysian and Singapore Food Composition Databases. The modified version of HEI used in this study consists of 14 components. Sum scores of each component yields and overall score of diet quality which will be converted into scale of zero to 100. A higher the HEI score indicates a greater adherence. The overall dietary adherence will be classified as low (below 51%), needing improvement (51-80%), or high (more than 80 points)

SECONDARY OUTCOMES:
Comparison of glycated hemoglobin (HbA1c) at 3-month and 6-month between the usual care group and intervention group | Baseline, 3-month, and 6-month
  Change in HbA1c will be determined by blood test at baseline, 3 and 6 months. The HbA1c result will be retrieved from the participants' routine blood result at health clinic or hospital, which will be analyzed following a standardized analytic protocol of Ministry of Health, Malaysia
Comparison of self-management behavior at 3-month and 6-month between the usual care group and intervention group | Baseline, 3-month, and 6-month
  The Malay version of the Summary of Diabetes Self-Care Activities (SDSCA) will be used to measure diabetes self-management activities. The SDSCA will be used to examine the participants' compliance in performing five main self-care activities. The degree of compliance or frequency with which the person engages in each self-care behavior is considered when interpreting the SDSCA scores. Higher ratings across the board typically suggest better adherence and more active diabetes self-management.

CONTACTS AND LOCATIONS:
Locations (1):
- Ranau District Hospital and Klinik Kesihatan Kundasang, Kota Kinabalu, Sabah, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arora S, Peters AL, Burner E, Lam CN, Menchine M. Trial to examine text message-based mHealth in emergency department patients with diabetes (TExT-MED): a randomized controlled trial. Ann Emerg Med. 2014 Jun;63(6):745-54.e6. doi: 10.1016/j.annemergmed.2013.10.012. Epub 2013 Nov 11. PMID 24225332
- [Background] Ramachandran A, Snehalatha C, Ram J, Selvam S, Simon M, Nanditha A, Shetty AS, Godsland IF, Chaturvedi N, Majeed A, Oliver N, Toumazou C, Alberti KG, Johnston DG. Effectiveness of mobile phone messaging in prevention of type 2 diabetes by lifestyle modification in men in India: a prospective, parallel-group, randomised controlled trial. Lancet Diabetes Endocrinol. 2013 Nov;1(3):191-8. doi: 10.1016/S2213-8587(13)70067-6. Epub 2013 Sep 11. PMID 24622367